CLINICAL TRIAL: NCT06589440
Title: Phase 2 Study of SR-8541A in Combination With Botensilimab and Balstilimab in Subjects With Refractory Metastatic Microsatellite Stable Colorectal Cancer (MSS-CRC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stingray Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR-8541A-002
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Refractory Metastatic Microsatellite Stable Colorectal Cancer (MSS-CRC)
MeSH Terms: interventions — balstilimab

STUDY DESIGN:
Intervention Model Description: Part 1 will follow a traditional 3+3 dose escalation scheme. Approximately 6-12 subjects will be treated in Part 1.
  Part 2 Approximately up to 58 subjects will be enrolled:
  Cohort A: MSS-CRC subject with no active liver metastases Cohort B: MSS-CRC subject with active liver metastases
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSS-CRC subject with no active liver metastases (Experimental)
  Interventions: Drug: SR-8541A
- MSS-CRC subject with active liver metastases (Experimental)
  Interventions: Drug: SR-8541A

INTERVENTIONS:
Drug: SR-8541A — SR-8541A administered orally in combination with intravenous botensilimab and balstilimab
  Other Names: Botensilimab; Balstilimab

SUMMARY:
This is an open-label, dose escalation and expansion, multi-center phase 2 study evaluating the safety and efficacy of SR-8541A administered orally in combination with intravenous botensilimab and balstilimab in subjects with MSS-CRC with and without active liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from subject
2. Age ≥ 18 years old on the date of consent
3. Histologically confirmed diagnosis of unresectable and metastatic adenocarcinoma of the colon or rectum
4. Non-microsatellite instability high or non-deficient mismatch repair (non-MSI-H/non-dMMR) tumor status per a standard local testing method
5. Must have received at least 1 prior chemotherapy regimen for metastatic or recurrent CRC
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Measurable disease per RECIST v1.1 (Eisenhauer et al., 2009)
8. Able to provide archival or fresh tumor tissue during screening (required) and post-treatment (optional)
9. Adequate renal function defined as creatinine clearance ≥ 60mL/min
10. Adequate liver function
11. Adequate hematologic function
12. No growth factor support, transfusions, or albumin administration within 14 days of first dose of study treatment
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
14. Male and female subjects of childbearing potential must agree to use a highly medically effective method of contraception and refrain from sperm/egg donation throughout the study starting with the first dose of study treatment (or 14 days prior to the first dose of study treatment for oral contraception) and for at least 3 months after the last dose of study treatment

Exclusion Criteria:

1. Hypersensitivity or allergy to any of the study drugs or their excipients.
2. In Part 2, Cohort A, active liver metastases by computed topography (CT) or magnetic resonance imaging (MRI).
3. Treatment with one of the following classes of drugs within the delineated time window prior to first dose:

   1. Small molecule/tyrosine kinase inhibitors within 2 weeks
   2. Any other systemic therapy for CRC within 3 weeks
   3. Received another investigational drug within 30 days or active participation in another clinical trial (follow-up is permitted)
   4. Medications/products which are known strong inhibitors or inducers of the CYP enzymes within 5 x T1/2
4. Received programmed cell death protein 1, PD-(L)1, or CTLA-4 therapies including any immune checkpoint inhibitor or experimental immunologic agents.
5. Partial or complete bowel obstruction within the last 3 months, signs/symptoms of bowel obstruction, or known radiologic evidence of impending obstruction.
6. Refractory ascites.
7. Current evidence of interstitial lung disease (ILD) or pneumonitis, or prior history of ILD or non-infectious pneumonitis requiring glucocorticoids.
8. Continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 28 days prior to Day 1.
9. Active autoimmune disease that has required systemic treatment in past 2 years
10. Patients with adrenal / pituitary insufficiency
11. History of documented congestive heart failure; unstable angina; poorly controlled hypertension; clinically significant valvular heart disease; high-risk uncontrolled arrhythmias (including sustained ventricular tachycardia); myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack within the last 6 months, or Canadian Cardiovascular Society angina class > 2
12. History of allogeneic organ transplant, stem cell transplant, or bone marrow transplant
13. Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to first dose
14. Requirement for treatment with strong cytochrome P450 3A4 inducers or inhibitors
15. Presence of gastrointestinal condition, for example, malabsorption, that might affect the absorption of Investigational Product(s).
16. Troponin I > ULN
17. Uncontrolled hypertension
18. Corrected QT interval by Fridericia (QTcF) ≥ 470 ms per the central mean average of triplicate electrocardiograms (ECGs)
19. Left Ventricular Ejection Fraction (LVEF) < 50% using echocardiogram or multigated acquisition (MUGA)
20. Symptomatic uncontrolled central nervous system (CNS) disease requiring treatment with steroids or anti-seizure medications within 2 months prior to Day 1. However, subjects with brain metastases that have been previously treated and are stable based on imaging performed within 2 months of Day 1 following completion of any CNS-directed therapy are allowed
21. Leptomeningeal disease
22. Spinal cord compression not definitively treated with surgery and/or radiation
23. Bleeding diathesis due to underlying medical condition or anticoagulation medication which is unable to be promptly reversed by medical treatment
24. Prior additional malignancy that is progressing or has received treatment the previous 3 years prior to first dose except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
25. History of uncontrolled seizures, central nervous disorders, substance abuse disorder or psychiatric disability judged by the Investigator to be clinically significant and would interfere with cooperation with requirements of the study
26. Active infection requiring systemic treatment at time of first dose
27. Positive for human immunodeficiency virus (HIV) (HIV antibodies) or active hepatitis B (e.g., HbsAg reactive) or active hepatitis C (e.g., HCV ribonucleic acid [RNA] qualitative) infection with detectable viral load
28. Pregnant or lactating females who plan to nurse a child during or within 3 months of the last dose of study treatment
29. Major surgery within 28 days prior to first dose and/or minor surgery (excluding biopsy) within 7 days prior to first dose. Note: If the subject had major surgery, the subject must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention
30. Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the subject or impair the assessment of study results
31. Planned use of any of the prohibited concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, efficacy, and define the optimal dose for expansion of SR-8541A in combination with botensilimab and balstilimab | Approximately 3 dose levels (DL) will be investigated in 28-day cycles
  Part 1 of the study is to establish the recommended dose of SR-8541A in combination with botensilimab and balstilimab.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Atlantic Health, Morristown, New Jersey
  - Texas Oncology- Austin, Austin, Texas
  - Texas Oncology- Sammons- DFW, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center GI Medical Oncology Dept, Houston, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
  - Swedish, Seattle, Washington